CLINICAL TRIAL: NCT00047073
Title: A Modified Phase I/II Trial Of Rapamycin In Patients With Glioblastoma Multiforme
Brief Title: Sirolimus in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Timothy Cloughesy, M.D., UCLA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257255; UCLA-0203078; NCI-G02-2114
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Sirolimus; Surgical Procedures, Operative; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 (Experimental): See intervention description.
  Interventions: Drug: Rapamycin; Procedure: Surgery; Procedure: Supportive Care
- Phase 2 (Experimental): See intervention description.
  Interventions: Drug: Rapamycin; Procedure: Surgery; Procedure: Supportive Care

INTERVENTIONS:
Drug: Rapamycin — Phase 1: Initial dose 6mg on day 1 and then 2mg each day for 5-7 days before surgery. No dosing during surgery recovery. After recorvery 6mg loading dose on day 1 then 2mg each day. Cycle is every 4 weeks.
  Dose escalation: Level 2: 15mg load/5mg/day, Level 3: 30mg load/10mg/day, Level 4: 45mg load/15mg/day.
  Phase 2: Will utilize dose established in phase I. Dosing schedule will remain the same.
  Other Names: Sirolimus
Procedure: Surgery — Surgical resection.
Procedure: Supportive Care — Corticosteroids should be used in smallest dose to control symptoms of cerebral edema and mass effect.
  Anti-seizure medications should be used as indicated. Febrile neutropenia may be managed according to local institution's infectious disease guidelines.
  If neurosurgical management is required for reasons not due to tumor progression, these procedures must be documented.

SUMMARY:
RATIONALE: Chemotherapy drugs such as sirolimus use different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase I/II trial to study the effectiveness of sirolimus in treating patients who have glioblastoma multiforme that did not respond to previous radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of sirolimus in patients with glioblastoma multiforme.
* Determine the safety profile of this drug in these patients.
* Determine the efficacy of this drug, in terms of 6-month progression-free survival and objective response, in these patients.

OUTLINE: This is a dose-escalation study.

* Phase I: Patients receive oral sirolimus for 5-7 days before surgery. Patients then undergo surgical resection. Patients resume oral sirolimus once daily after full recovery from surgery. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of sirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive oral sirolimus as in phase I at the dose determined in that phase.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 3-12 patients will be accrued for phase I of the study within 3-12 months. A total of 32 patients will be accrued for phase II of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial glioblastoma multiforme
* Disease progression by MRI or CT scan

  * Confirmation of true progressive disease (not radiation necrosis) by positron-emission tomography, thallium scanning, MRI, or surgical documentation required if patient received prior interstitial brachytherapy or stereotactic radiosurgery
* Failed prior radiotherapy
* Phase I patients:

  * Eligible for salvage surgery
  * No limits on prior therapy
* Phase II patients:

  * Tumor progression by MRI or CT scan required within the past 14 days if recurrent disease is present
  * No prior therapy for more than 3 relapses
  * Recent resection of recurrent or progressive tumor allowed as long as all of the following conditions apply:

    * Recovered from surgery
    * MRI or CT scan performed no more than 96 hours since prior surgery OR within 4-6 weeks after surgery
    * Baseline MRI or CT scan performed within 14 days of study entry

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT less than 1.5 times ULN

Renal

* Creatinine less than 1.5 mg/dL

Other

* Cholesterol less than 350 mg/dL
* Triglycerides less than 400 mg/dL
* No concurrent disease that would obscure toxicity or dangerously alter drug metabolism
* No other significant uncontrolled serious medical illness that would preclude study participation
* No other cancer except non-melanoma skin cancer or carcinoma in situ of the cervix unless patient is in complete remission and off all therapy for that disease for at least 3 years
* No active infection
* No prior allergic reactions to compounds of similar chemical or biological composition to sirolimus
* No psychiatric illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 1 week since prior interferon

Chemotherapy

* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 6 weeks since prior nitrosoureas

Endocrine therapy

* At least 1 week since prior tamoxifen

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* Recovered from prior therapy
* At least 1 week since prior noncytotoxic agents (except radiosensitizers)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-07; Primary Completion 2005-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (for phase 1) | end of phase 1
Efficacy in terms of progression-free survival at 6 months and objective response (phase II) | 6 months after last subject finishes trial

SECONDARY OUTCOMES:
Safety Profile (phase I) | end of phase I
Further evaluate safety profile | end of phase II

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F. Cloughesy, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Cloughesy TF, Yoshimoto K, Nghiemphu P, Brown K, Dang J, Zhu S, Hsueh T, Chen Y, Wang W, Youngkin D, Liau L, Martin N, Becker D, Bergsneider M, Lai A, Green R, Oglesby T, Koleto M, Trent J, Horvath S, Mischel PS, Mellinghoff IK, Sawyers CL. Antitumor activity of rapamycin in a Phase I trial for patients with recurrent PTEN-deficient glioblastoma. PLoS Med. 2008 Jan 22;5(1):e8. doi: 10.1371/journal.pmed.0050008. PMID 18215105